CLINICAL TRIAL: NCT07090785
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY4088044 in Healthy Participants.
Brief Title: A Study of LY4088044 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27275; J5S-MC-CEAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-07-09; First posted 2025-07-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY4088044 (Part A) (Experimental): Single-ascending dose (SAD) of LY4088044 administered intravenously (IV)
  Interventions: Drug: LY4088044
- Placebo (Part A) (Placebo Comparator): Administered IV
  Interventions: Drug: Placebo
- LY4088044 (Part B) (Experimental): SAD of LY4088044 administered subcutaneously (SC)
  Interventions: Drug: LY4088044
- Placebo (Part B) (Placebo Comparator): Administered SC
  Interventions: Drug: Placebo
- LY4088044 (Part C) (Experimental): Multiple-ascending doses (MAD) of LY4088044 administered IV
  Interventions: Drug: LY4088044
- Placebo (Part C) (Placebo Comparator): Administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4088044 — Administered IV
  Arms: LY4088044 (Part A); LY4088044 (Part C)
Drug: LY4088044 — Administered SC
  Arms: LY4088044 (Part B)
Drug: Placebo — Administered IV
  Arms: Placebo (Part A); Placebo (Part C)
Drug: Placebo — Administered SC
  Arms: Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate how well LY4088044 is tolerated and what side effects may occur in healthy participants. The study drug will be administered either subcutaneously (SC) (under the skin) or intravenously (IV) (into a vein in the arm). Blood tests will be performed to check how much LY4088044 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 92 weeks for Parts A, B, and C, excluding screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and cardiac monitoring
* Have a body mass index (BMI) within the range 18.5 to 30 kilogram per square meter (kg/m²)

Exclusion Criteria:

* Are individuals assigned female at birth (AFAB) who are pregnant and/or lactating
* Regularly use known drugs of abuse or show positive findings on urinary drug screening that are not consistent with their medication history
* Participants with hemoglobin outside of the local laboratory normal range for age and gender, or evidence of iron deficiency, or hemoglobinopathy
* Participants with estimated glomerular filtration rate (GFR) less than 90 milliliter per minute per 1.73 square meter (mL/min/1.73 m²)
* Have a 12-lead electrocardiogram (ECG) abnormality
* Smoke more than 10 cigarettes per day or the equivalent including electronic cigarettes AND are unable to abide by investigative site smoking restrictions
* Have an average weekly alcohol intake that exceeds 21 units per week (males less than or equal to 65 years old) and 14 units per week (females and males over 65-year-old, if applicable) and are unwilling to abide by the restrictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Day 190
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4088044 | Baseline up to Approximately Day 190
  PK: Cmax of LY4088044
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4088044 | Baseline up to Approximately Day 190
  PK: AUC of LY4088044
Pharmacodynamics (PD): Protein Levels in Skin Samples | Baseline up to Approximately Day 190
  PD: Percent Decrease in Protein Levels

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (4):
  - Collaborative Neuroscience Network - CNS, Los Alamitos, California
  - ICON, Lenexa, Kansas
  - ICON Early Phase Services, San Antonio, Texas
  - ICON, Salt Lake City, Utah
- New Zealand Clinical Research Christchurch, Christchurch, New Zealand
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No